CLINICAL TRIAL: NCT02044016
Title: The Achilles Tendon Length Measure (ATLM) - Development and Validation
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Maria Swennergren Hansen, Physiotherapist, Hvidovre University Hospital
Other Study IDs: H-4-2013-FSP
Record Dates: First submitted 2014-01-20; First posted 2014-01-23 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Achilles Tendon Rupture
Keywords: Achilles tendon rupture, lengthening, validity, goniometer.

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational study: To compare results of the ATLM with goniometry and Ultrasound measures of the achilles tendon.

SUMMARY:
The purpose of this study is 1) to develop and validate a new measurement to assess the length of the Achilles tendon after rupture, and 2) to examine if goniometer measurement of the ankle joint is a better method.

DETAILED DESCRIPTION:
It has been shown that an Achilles tendon elongation compared to the un-injured leg is negatively associated with the clinical outcome and strength of the gastrocnemius muscle. Despite this knowledge, there is a lack of a valid score system that can measure the length of the Achilles tendon in daily clinical practice. Patients, who follow a rehabilitation program at the Department of Physiotherapy, also have their Achilles tendon examined for lengthening by physiotherapists, to evaluate if the heeling progresses as planned. Of concern, this examination is based on measures, which have not been thoroughly validated.

The ATLM test use the same test position of the lower limb as being used in Matles test. Besides observing the foot's position, we will measure the distance from a point of reference on the foot to the examination coach. Reproducibility and responsiveness of the ATLM will be examined, while concurrent validity will be examined against ultrasound and a goniometry measure. The ultrasound is considered the most precise, secure and objective measure.

The ATLM and goniometer measures will be conducted at 8 and 16 weeks after the injury. At 8 weeks there will be two physiotherapists conducting these measures (to investigate inter-tester reliability). The ruler and goniometer will have the numbers hidden. A third physiotherapist will read the results at 8 and 16 weeks, so that the physiotherapists will be blinded towards the results. A person blinded to these results will conduct the ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-60.
* Patients who are being referred to the rehabilitation program for patients with an AATR, at Hvidovre Hospital.
* The patients have to speak and understand Danish.
* The patients have to be able to sign the written informed consent.

Exclusion Criteria:

* Patients who earlier have had a rupture of one or both AT.
* Patients who have had an operation one of the achilles tendons before.
* Patients who have been diagnosed with arterial insufficiency in legs.
* Patients with a terminal disease or who suffers from a critical medical illness.
* Patients where the distance from rupture to calcaneus is less than 1 cm (examined by palpation or in doubt, measured with an ultrasound)
* Fluoroquinolone treatment within the last 6 months.
* Tendinosis treated with corticosteroids (tablets or injections) within the last 6 months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with an acute achilles tendon rupture, between week 8 and 16 after injury. The patients are participating in a rehabilitation exercise group led by a physiotherapist 2 times a week for one hour at the time. Therefore, the patients in this study will be recruited from this program, and if they accept, they will be followed through the program, during the 2 examinations.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2014-04; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Achilles Tendon Length Measure (ATLM) | 8 weeks after injury
  The tester position one leg with a knee joint ankle to 90 degrees flexion. The other hand of the tester holds the ruler op against the foot. A plate in a hard, stiff wooden material is placed underneath the patient's thighs and knees. A ruler that is 100 cm long (25x5 mm) made in wood is being used. The tester is seated at the end of the examination coach. Besides observing the foot's position, we will measure the distances from points of reference on the foot to the examination coach. Points of reference: 1) The middle (and most prominent) point of the head of the fifth metatarsophalangeal head seen from the lateral side. 2) From the middle point of the lateral malleolus down to the examination coach).Take the first measure (metatarsophalangeal head-examination coach) and subtract this with the second one (lateral malleolus-examination coach). See if there is a difference between uninjured and injured side. Here you get the ATLM.

SECONDARY OUTCOMES:
Goniometer measurement of the angle in the ankle joint | 8 weeks after injury
  Position of the subject is prone with the knee on the testing side being tested flexed to 90 degrees. The patients is is being encouraged to relax as much as possible. Centre fulcrum of the goniometer over the lateral aspect of the lateral malleolus. The proximal arm of the goniometer with the lateral midline of the fibula, using the head of the fibula for reference. The distal arm of the goniometer parallel to the lateral aspect of the fifth metatarsal. The relaxed position of the ankle is being measured.
Ultrasound | 8 weeks after injury
  The patient is lying on the stomach with the knees slightly bent and ankle joints in about 15-20 degrees of plantar flexion. Two points of reference is being marked with a single dot by a pencil: 1. The proximal part of calcaneus. The ultrasound-probe is being oriented in the length of the shank. The most proximal spot of calcaneus is being localised. With a needle under the probe (upon the skin), there is a spot on the skin where the shadow spots a place where corticalis on calcaneus is being forfeit in the depth. 2. The distal tip of the medial head of the gastrocnemius. The ultrasound-probe is being oriented of the length of the shank. With a needle under the probe (upon the skin) a place on the skin exists, where the shadow spots the distal peak of the medial gastrocnemius head. The distance between the marks is being measured outside the skin with a tapeline following the contour of the shank.
Goniometer measurement of the angle in the ankle joint | 16 weeks after injury
  The same test as after 8 weeks.
Ultrasound | 16 weeks after injury
  The same test as after 8 weeks.
Achilles Tendon Length Measure (ATLM) | 16 weeks after injury
  The same test as after 8 weeks.

OTHER OUTCOMES:
Achilles tendon Total Rupture Score | A couple of days after date of injury
  A patient reported validation score developed to assess symptoms and physical activity after treatment for Achilles tendon rupture.
Heel-rise work test | 16 weeks after injury.
  Endurance test where the patient stands on one leg and lifts the heel up and down until exhaustion. The number and the height of the heel-rises are counted and measured. The results are then compared to the weight of the patient and the total work is estimated. The MuscleLab ® (Ergo Test Technology, Oslo, Norway) measurement system is used.
Heel-rise height test | 16 weeks after injury
  The patient stands facing a wall. The patient is allowed to hold 3 fingers on each hand up against the wall for support. The patient is asked to first stand on the un-injured leg and rise the heel as far up as possible. The distance between the calcaneus and the floor is being measured in millimeters. The same procedure is there after performed on the injured leg.
Physical Activity Scale (PAS) | A couple of days after date of injury
  The PAS is an instrument that measures the level of physical activity among adults.
Achilles tendon Total Rupture Score | 16 weeks after injury
  The same as after 8 weeks.
Physical Activity Scale (PAS) | 16 weeks after injury
  The same as after 8 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Svennergren, Principal Investigator — Hvidovre University Hospital Denmark, Department of Physiotherapy
Locations (1):
- Department of Physiotherapy, Hvidovre University Hospital, Copenhagen, Hvidovre, Denmark